CLINICAL TRIAL: NCT00943605
Title: A Prospective, Randomized, Controlled Superiority Study to Evaluate Use of the PEAK PlasmaBlade™ 4.0 in Mastectomy
Brief Title: PEAK PlasmaBlade™ 4.0 Versus Traditional Electrosurgery in Mastectomy
Acronym: PRECISE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Termination due to acquisition of PEAK Surgical by Medtronic
Sponsor: Medtronic Surgical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PEAK VP-00074
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Results first posted 2013-01-03 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Mastectomy
Keywords: Mastectomy; PlasmaBlade; Electrosurgery; PEAK Surgical; Medtronic Advanced Energy; Medtronic
MeSH Terms: conditions — Hyperthermia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (Active Comparator): Scalpel will be used for the skin incision and traditional electrosurgery for the subcutaneous dissection.
  Interventions: Device: Scalpel and Traditional Electrosurgery
- PEAK PlasmaBlade (Experimental): The entirety of the mastectomy will be performed with the PEAK PlasmaBlade, including the skin incision.
  Interventions: Device: PEAK PlasmaBlade

INTERVENTIONS:
Device: Scalpel and Traditional Electrosurgery — The PEAK PlasmaBlade will be used for the entirety of the breast reduction, including the skin incision.
  Arms: Standard of Care
Device: PEAK PlasmaBlade — The entirety of the mastectomy will be performed with the PEAK PlasmaBlade, including the skin incision.
  Arms: PEAK PlasmaBlade

SUMMARY:
The objective of this clinical study is to evaluate the incidence of partial skin necrosis following modified-radical mastectomy with or without same-day (two-stage) reconstruction with the PEAK PlasmaBlade 4.0; to monitor and record operative performance, post-operative pain, drain output, and skin scarring following surgery; and to compare these endpoints to the current standard of care (SOC).

DETAILED DESCRIPTION:
Mastectomy is a surgical procedure performed to remove breast tissue that contains cancer, or has a high probability of containing cancer. During the procedure, a scalpel is used for the skin incision and a traditional electrosurgical device is used to cut away the breast tissue from the chest and control bleeding. Once the breast tissue is removed the remaining skin edges are brought together with sutures.

Following mastectomy, the most common complication is persistent serous wound drainage and seroma, a collection of fluid in the closed surgical space. To help prevent this complication a tissue drain is used to remove serous fluid from the surgical space via bulb suction. The rate of serous fluid collection is used to determine the time the drain remains in place. Although suction drains help reduce seroma formation, prolonged use may delay healing, cause injury, and increase the risk of infection and patient discomfort.

The PEAK PlasmaBlade™ uses pulsed radiofrequency (RF) energy to enable precision cutting and coagulating at the point of application, without the thermal damage to surrounding tissues that is normally seen with traditional electrosurgery. The PlasmaBlade has received FDA clearance for use in plastic, general, and ENT surgery, and has demonstrated significantly reduced serous drainage in tissue reduction surgeries, like mastectomy.

This multi-site study was granted IRB approval and conducted between June 2009 and January 2011. Potential subjects were screened against the inclusion and exclusion criteria of the study protocol and were then required to provide informed consent prior to enrollment. Following enrollment, subjects were prospectively randomized to the SOC or PlasmaBlade (PB or PEAK) study groups and scheduled for mastectomy with or without same day reconstruction.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20 and 70 years old
2. Physically healthy, stable weight
3. Requiring single or bilateral simple mastectomy, with or without sentinel lymph node biopsy
4. Subject must understand the nature of the procedure and provide written informed consent prior to the procedure
5. Subject must be willing and able to comply with all follow-up evaluations

Exclusion Criteria:

1. Age younger than 20 or greater than 70 years old
2. Anticoagulation therapy which cannot be discontinued
3. Prior external beam or implanted radiotherapy
4. Tobacco use (any kind)
5. Infection (local or systemic)
6. Cognitive impairment or mental illness
7. Severe cardiopulmonary deficiencies
8. Known coagulopathy
9. Immunocompromised
10. Kidney disease (any type)
11. Desiring or requiring same-day breast reconstruction
12. Prior breast reduction or augmentation surgery
13. Unable to follow instructions or complete follow-up
14. Currently taking any medication known to affect healing
15. Subjects who are status-post gastric banding or gastric bypass
16. Currently enrolled in another investigational device or drug trial
17. Time from most recent neoadjuvant therapy less than 4 weeks

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-06; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Ponn, MD, Principal Investigator — Elliot Breast Health Center; Edward Dalton, MD, Principal Investigator — Elliot Breast Health Center; Richard Fine, MD, Principal Investigator — Advanced Breast Care; Peter Naruns, MD, Principal Investigator — Midpeninsula Surgical Associates; Saul Eisenstat, MD, Principal Investigator — Midpeninsula Surgical Associates; Michael Schultz, MD, Principal Investigator — St. Joseph Medical Center
Locations (4):
- United States (4):
  - Providence St. Joseph's Medical Center, Burbank, California
  - El Camino Hospital, Mountain View, California
  - Advanced Breast Care, Marietta, Georgia
  - St. Joseph Medical Center, Towson, Maryland

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care (SOC): Scalpel will be used for the skin incision and traditional electrosurgery for the subcutaneous dissection.
Period: Overall Study
Arm/Group | Standard of Care (SOC) | PEAK PlasmaBlade
Started | 30 (There were 10 total subjects (5/group) who were retrospectively unenrolled for deviations.) | 30 (There were 10 total subjects (5/group) who were retrospectively unenrolled for deviations.)
Completed | 0 | 0
Not Completed | 30 | 30
Not completed — Study termination | 30 | 30

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care (SOC) | PEAK PlasmaBlade | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Customized [Number; unit: participants] — An integrity audit found that the data for this study could not be analyzed owing to unverifiable source documentation. The protocol-specified age range is used for this baseline measure.
  participants
    20 to 70 years | 30 | 30 | 60
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Total Serous Drainage (mL) From Time of Drain Placement to Removal.
Time Frame: 0 to 10 days postoperatively
Population: An integrity audit found that the data for this study could not be analyzed owing to unverifiable source documentation.
Arm/Group | Standard of Care (SOC) | PEAK PlasmaBlade
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Area of Skin Necrosis Measured With a Standard Ruler
Time Frame: 1 and 6 weeks postoperative
Population: An integrity audit found that the data for this study could not be analyzed owing to unverifiable source documentation.
Arm/Group | Standard of Care (SOC) | PEAK PlasmaBlade
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Pain Score by Visual Analog Scale, Narcotic Consumption, Operative Time, Time to Surgical Drain Removal
Time Frame: 0 to 10 days postoperatively
Population: An integrity audit found that the data for this study could not be analyzed owing to unverifiable source documentation.
Arm/Group | Standard of Care (SOC) | PEAK PlasmaBlade
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Standard of Care (SOC) | PEAK PlasmaBlade
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 4/30 | 2/30
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (SOC) (N=30) | PEAK PlasmaBlade (N=30)
Seroma (Surgical and medical procedures) | 2 (2) | 1 (1)
Fluid aspiration (Surgical and medical procedures) | 1 (1) | 1 (1)
Incision opened and resutured (Surgical and medical procedures) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Upon Medtronic's acquisition of PEAK surgical, a study integrity audit was undertaken. Results of the audit showed that patient's rights and safety were maintained, but the source data, including baseline demographics, were unverifiable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less